CLINICAL TRIAL: NCT02817412
Title: Food Response Training for Binge Eating
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principle investigator (Sylvia Herbozo) left the university.
Sponsor: Loma Linda University (Other)
Collaborators: Oregon Research Institute (Other)
Responsible Party: Principal Investigator, Holly Morrell, Associate Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5160020
Record Dates: First submitted 2016-06-23; First posted 2016-06-29 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Binge Eating
Keywords: binge eating; obesity; overeating
MeSH Terms: conditions — Bulimia; Obesity; Hyperphagia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Go/No-Go Training (Experimental): In the go/no go training, participants are shown images in which high-calorie foods are shown on one side of the screen and low-calorie foods on the other. They are told to press response keys as quickly as possible to indicate the side of presentation (go-trials). On half of the trials, the rectangular frame surrounding the image is not solid but hatched, which is a signal for them to withhold their response (no-go trials). This training is divided into 4 blocks of 50 trials.
  Interventions: Behavioral: Go/No-Training
- Stop-Signal Training (Experimental): In the stop signal training, participants are shown images in either a dark blue or light gray border. They are told to press the space bar as quickly as possible when the border is blue (go trials) and to withhold a response when the border is gray (no-go trials). This training is divided into 20 blocks of 32 trials.
  Interventions: Behavioral: Stop-Signal Training
- Dot-Probe Training (Experimental): In the dot-probe training, participants are shown images in which high-calorie foods are shown on one side of the screen and low-calorie foods on the other. Immediately after the images disappear, a small dot probe appears in the location of one of the images. Participants are told to press response keys as quickly as possible to indicate whether a visual probe appeared behind the left or right image during the trials. The probe appears in the location occupied by a high-calorie food image 10% of the time and in the location occupied by a low-calorie food image 90% of the time. This training is divided into 6 blocks of 40 trials.
  Interventions: Behavioral: Dot-Probe Paradigm
- Generic Training (Placebo Comparator): In the generic training, participants complete a generic go/no-go training that uses images of flowers and office supplies instead of the images of high-calorie and low-calorie food images. This generic go/no go training is identical in duration and contact time to the go/no-go food training.
  Interventions: Behavioral: Generic Response Training

INTERVENTIONS:
Behavioral: Go/No-Training
  Arms: Go/No-Go Training
Behavioral: Stop-Signal Training
  Arms: Stop-Signal Training
Behavioral: Dot-Probe Paradigm
  Arms: Dot-Probe Training
Behavioral: Generic Response Training
  Arms: Generic Training

SUMMARY:
This study will examine the effectiveness of food response training interventions in reducing binge eating among adults engaged in binge eating.

DETAILED DESCRIPTION:
Binge eating disorder is the most prevalent eating disorder and affects both men and women at comparable rates unlike anorexia nervosa and bulimia nervosa. Given that binge eating and obesity are strongly associated, binge eating treatments should aim to reduce binge eating as well as weight. However, most binge eating interventions do not produce lasting weight loss. Recent research has shown computer-based response inhibition training with high-calorie foods reduces reward region response to and attentional bias for the training foods, decreases training food intake, increases inhibitory control, and produces weight loss in overweight adults. There is evidence that the weight loss effects from such response training persist through 6-month follow-up. Further, binge eating has been associated with increased food-related impulsivity and increased activation in a reward-processing brain region to high-calorie foods. Prior research suggests that food response training may be an effective intervention for binge eating that teaches automatic self-control in response to high-calorie foods which in turn, reduces binge eating and produces weight loss. This study will examine the effectiveness of food response training interventions in reducing binge eating and weight among adults engaged in binge eating.

The goals of this study are to: (1) test the hypothesis that adults who complete the food response trainings will show significantly greater reductions in binge eating frequency and in body mass index (BMI) compared to generic response training from pretest to posttest and at 3-month follow up, (2) to determine whether one of the food response trainings is more effective in binge eating frequency and reducing BMI from pretest to posttest and at 3-month follow up, and (3) test whether a reduction in valuation of the high-calorie versus low-calorie foods (willingness to pay for the pictured foods) and/or behavioral improvement of inhibitory control during the training tasks mediate the effects of the various trainings on reductions in binge frequency and body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Engages in objective binge episodes as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and meets one of the following frequency and duration criteria: 1) at least two objective binge episodes per month for at least 3 months; or 3) at least six objective binge episodes over a shorter period

Exclusion Criteria:

* Illicit drug use and excessive alcohol use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Binge Eating Frequency | Post-intervention (at 4 months)
  Number of times engaged in binge eating (self-report)
Binge Eating Frequency | 3-month follow-up (at 7 months)
  Number of times engaged in binge eating (self-report)

SECONDARY OUTCOMES:
Body Mass Index | Post-intervention (at 4 months)
  Weight in kilograms divided by height in meters squared.
Body Mass Index | 3-month follow-up (at 7 months)
  Weight in kilograms divided by height in meters squared.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Herbozo, Ph.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- Sylvia Herbozo, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No